CLINICAL TRIAL: NCT01523197
Title: Effect of Auto-Trilevel Ventilation on Patients With Overlap Syndrome
Brief Title: Auto-trilevel Ventilator for Patients With Overlap Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhang Xilong, Department of Respirology, The First Affiliated Hospital of Nanjing Medical University, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CXZZ11-0711
Record Dates: First submitted 2012-01-12; First posted 2012-02-01 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Overlap Syndrome
Keywords: Obstructive Sleep Apnea hypopnea Syndrome; COPD; overlap syndrome; Auto-trilevel ventilation; BiPAP ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ventilator (Other): The comparison of the curative effect on OS between BiPAP and auto-trilevel ventilations
  Interventions: Device: BiPAP ventilation, auto-trilevel ventilation

INTERVENTIONS:
Device: BiPAP ventilation, auto-trilevel ventilation — Noninvasive ventilation including fixed BiPAP ventilation and auto-trilevel ventilation. Using the same IPAP, treatment include one night with BiPAP ventilation mode 1, one night with BiPAP ventilation mode 2 and one night with auto-trilevel ventilation mode. Each treatment last 8 hours for each night.
  Other Names: bi-level postive airway preesure ventilation;; auto-trilevel ventilation

SUMMARY:
Obstructive Sleep Apnea Syndrome (OSAS) and chronic obstructive pulmonary disease (COPD) are two diseases that often coexist and are called overlap syndrome(OS). Compared to single OSAS, OS patients are more susceptible to serious hypoxia and hypercapnia especially during sleep, and are much more likely to result in pulmonary hypertension and cor-pulmonal.

With a more flexible expiratory positive airway pressure (EPAP), auto-trilevel ventilation may be superior to fixed bilevel positive airway pressure (BiPAP) ventilation in both removing residual obstructive sleep apnea hypopnea events and correcting hypercapnia simultaneously. The overall purpose of this study is to compare the curative effects between fixed BiPAP and auto-trilevel ventilations on OS patients.

DETAILED DESCRIPTION:
The contradiction in treatment for overlap syndrome is how to improve hypercapnia because of narrower difference between inspiratory positive airway pressure (IPAP) and expiratory positive airway pressure (EPAP), and meanwhile to eliminate apnea and popnea events which may easily occur at the end of expiration For ordinary Bipap ventilator. If the IPAP is set to higher, the patients may feel discomfort, if the pressure difference between IPAP and EPAP is too narrow or the expiratory positive airway pressure (EPAP) too high, hypercapnia may occur. If the EPAP is too low, redusual apnea and hypopnea event may become common.

Auto-trilevel ventilation, with a lower airway pressure at the beginning of expiration to prevent hypercapnia and a higher airway pressure at the end of expiration to prevent residual apnea events, should be able to provide a novel ventilation mode with a higher efficacy and lower average airway pressure for overlap syndrome. To prove the hypothesis, comparison is made between ordinary BiPAP and auto-Trilevel ventilation modes during treatment for patients with overlap syndrome.

In this study, the investigators compare the changes of related indexes including apnea hypopnea index、minimal pulse oxygen saturation、arousal index, sleep quality,PaCO2 and sleepiness scores) before and on treatment. Meanwhile, curative effects will be compared between BiPAP and auto-Trilevel ventilation modes. The investigators will analyze the changes and then confirm our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legal representative of the patient is willing and able to sign an approved informed consent and privacy protection authorization in the United States.
2. Subject is >18 years old.
3. Diagnosed overlap syndrome(OSAS and COPD). 4. Expected to tolerate the ventilator therapy .

Exclusion Criteria:

1. Patient is currently enrolled in another clinical study which may confound the result of this study.
2. Patient for who inform consent cannot be obtained.
3. Patients with a history of cerebrovascular accident within the 6 months prior to this study.
4. Patients with acute or chronic renal failure, diabetes and severe lung diseases.
5. Patients with unstable angina.
6. Patient who is of pregnant or during lactation period.
7. Patients with a history of injury or surgery within 6 months prior to the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
different effects between BiPAP and auto-Trilevel ventilators on OS | Participants will be observed for the duration of hospital stay, an expected average of 1 weeks
  The overall purpose of this study is to determine the effects of auto-Trilevel ventilation on patients with overlap syndrome by comparison with BiPAP ventilation. The following parameters are compared such as apnea hypopnea index, lowest SPO2, arousal index, sleep efficiency, PaCO2, daytime sleepiness and so on.

CONTACTS AND LOCATIONS:
Overall Officials: xilong zhang, MD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China